CLINICAL TRIAL: NCT05687045
Title: High-flow Nasal Cannula Oxygen Therapy for Outpatients Undergoing Colonoscopy: a Randomized Controlled Trial
Brief Title: High Flow Nasal Cannula in Patients Undergoing Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Colon-HFNC
Record Dates: First submitted 2022-11-14; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Colonoscopy
Keywords: colonoscopy; High Flow Nasal Cannula; Gas exchange

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Experimental): High Flow Nasal cannula is a system to deliver heated and humidified oxygen with an inspired oxygen fraction between 21 and 100% through large bore nasal cannula. The system delivers a flow up to 60 liters/min.
  Interventions: Device: High Flow Nasal Cannula
- Standard Treatment (Active Comparator): If peripheral oxygen saturation will be < 95%, conventional oxygen therapy will be administered through common nasal cannula with a flow up to 6 Liters per minute
  Interventions: Device: Conventional Oxygen Therapy

INTERVENTIONS:
Device: High Flow Nasal Cannula — High Flow Nasal Cannula will be set at 60 liters per minute of air/oxygen admixture to reach a peripheral oxygen saturation equal or greater than 94%
  Arms: High Flow Nasal Cannula
Device: Conventional Oxygen Therapy — Conventional Oxygen Therapy will be administered through nasal cannula with a oxygen flow set to achieve a peripheral oxygen saturation equal or greater than 94%
  Arms: Standard Treatment

SUMMARY:
During colonoscopy, the insertion of the fiberscope and colon distension required to perform the examination may induce modifications to respiratory mechanics, respiratory effort and breathing pattern.

High-flow nasal cannula (HFNC) therapy is a mixed air-oxygen supply system able to deliver heated humidified gas up to 60 L/min of flow rate, with an inspiratory oxygen fraction (FiO2) ranging from 21% to 100%. Increasing evidence supports the use of HFNC in several clinical conditions and settings. When compared to standard therapy (ST), HFNC results in enhanced gas exchange and improved comfort.

No studies have yet assessed the benefits of HFNC versus ST during and after colonoscopy. The investigators designed this unblinded randomized controlled trial to assess whether HFNC, compared to ST, improves oxygenation at the end of the procedure (primary endpoint). Additional endpoints were: 1) the lowest peripheral saturation of oxygen (SpO2) and the number of oxygen desaturations; 2) the changes of end-expiratory lung impedance and tidal impedance assessed by Electrical Impedance Tomography (EIT); 3) the effects on diaphragm function assessed by ultrasound (DUS).

ELIGIBILITY:
Inclusion Criteria:

* outpatients with the indication to diagnostic colonoscopy

Exclusion Criteria:

* life-threatening cardiac aritmia or acute miocardical infarction within 6 weeks
* need for invasive or non invasive ventilation
* presence of pneumothorax or pulmonary enphisema or bullae
* recent (within 1 week) thoracic surgery
* presence of chest burns
* presence of tracheostomy
* pregnancy
* nasal or nasopharyngeal diseases
* dementia
* lack of consent or its withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gases at end of the procedure | At the end of the endoscopy
  Arterial blood will be sample for gas analysis

SECONDARY OUTCOMES:
Respiratory effort at end of the procedure | At the end of the endoscopy
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort at baseline | At enrollment
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort at the beginning of the colonoscopy | At 5 minutes after the beginning of the procedure
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Respiratory effort after the colonoscopy | After 10 minute from the end of the endoscopy
  The respiratory effort will be assessed through the ultrasonographic assessment of the diaphragm thickening fraction
Change of end-expiratory lung impedance (dEELI) from baseline at the beginning of the colonoscopy | At 5 minutes after the beginning of the procedure
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline at end of the procedure | At the end of the endoscopy, compared to baseline
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Change of end-expiratory lung impedance (dEELI) from baseline after colonoscopy | After 10 minute from the end of the endoscopy, compared to baseline
  change from baseline, expressed in mL, of the end expiratory lung volume as assessed through electrical impedance tomography
Arterial blood gases at baseline | At enrollment
  Arterial blood will be sample for gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, Principal Investigator — Magna Graecia University
Locations (1):
- AOU Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
The full protocol, datasets used and analysed during the current study will be available on reasonable request e-mailing the corresponding author
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be shared after results publication of indexed journal in english language
Access Criteria: On reasonable request